CLINICAL TRIAL: NCT00205010
Title: Laparoscopic Sentinel Lymph Node Localization in Patients With Operable Cervical Cancer - A Pilot Study
Brief Title: Laparoscopic Sentinel Lymph Node Localization in Operable Cervix Cancer
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: CO03701; H-2003-0442 (Other: Institutional Review Board); A532820 (Other: UW Madison); SMPH/OBSTET & GYNECOL (Other: UW Madison)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2008-06

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Lymphoscintigraphy

SUMMARY:
The purpose of this study is to evaluate the feasibility, safety and efficacy of laparoscopic ovarian transposition in women less than 40 years of age with locally advanced cervical squamous cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Stage IAI to IIA cervix cancer undergoing primary surgical management

Exclusion Criteria:

* Previous pelvic dissection
* Previous para-aortic lymph node dissection
* Evidence of distant mets

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-10; Primary Completion 2006-02 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Kushner, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Result] Kushner DM, Connor JP, Wilson MA, Hafez GR, Chappell RJ, Stewart SL, Hartenbach EM. Laparoscopic sentinel lymph node mapping for cervix cancer--a detailed evaluation and time analysis. Gynecol Oncol. 2007 Sep;106(3):507-12. doi: 10.1016/j.ygyno.2007.04.031. Epub 2007 Jun 8. PMID 17560635
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu